CLINICAL TRIAL: NCT04825301
Title: Application of Machine Learning Based Approaches in Emergency Department to Support Clinical Decision Managing SARS-CoV-2 Infected Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Clara Balsano, Full Professor, University of L'Aquila
Other Study IDs: prot. N. 28958
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Covid19; machine learning; prediction model; convolutional neural network
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training cohort: data collection
- validation cohort: data collection

SUMMARY:
The aim of the study is to develop a prognostic prediction model based on machine learning algorithms in patients affected by coronavirus disease 2019 (COVID-19), the prediction model will be capable to recognize patient with favorable prognosis or patient with poor prognosis by intelligent systems data analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 18 positive for COVID-19 by polymerase chain reaction assay for rhino-pharyngeal swab

Exclusion Criteria:

* Under 18 aged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Italian caucasian patients aged over 18 years old SARS-CoV-2 infection confirmed by PCR
Sampling Method: Probability Sample
Enrollment: 779 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 clinical course | 2 months
  Data about sex, age, symptoms start date, symptoms, comorbidity, vital parameters, hematochemical blood tests, therapy, oxygen support, radiology, clinical disease progression will be collected. The collected data will be analyzed through a machine learning based approach to predict the prognosis of patients affected by COVID-19.

SECONDARY OUTCOMES:
Application of machine learning algorithms on data of patients affected by COVID-19 | 2 months
  The collected data will be analyzed through a machine learning based approach to establish correlations between collected data and the prognosis of patients affected by COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Italy